CLINICAL TRIAL: NCT04201249
Title: MILES STUDY - Mesotherapy In Lateral Epicondylitis, a Prospective Randomized Controlled Study
Brief Title: Mesotherapy In Lateral Epicondylitis
Acronym: MILES
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Vítor Teixeira, Vitor Teixeira, Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MILES
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Piroxicam; Lidocaine; Mesotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesotherapy with piroxicam and lidocaine (Active Comparator)
  Interventions: Drug: Piroxicam, lidocaine
- Mesotherapy without piroxicam and lidocaine (Sham Comparator)
  Interventions: Device: Mesotherapy without drug administration

INTERVENTIONS:
Drug: Piroxicam, lidocaine — Patients will be randomized to 2 groups group A - mesotherapy with piroxicam (20mg/ml, 1ml) and lidocaine (1%, 1.5ml) (treatment arm); group group B - mesotherapy without piroxicam
  Arms: Mesotherapy with piroxicam and lidocaine
Device: Mesotherapy without drug administration — Patients will be randomized to 2 groups group A - mesotherapy with piroxicam (20mg/ml, 1ml) and lidocaine (1%, 1.5ml) (treatment arm); group group B - mesotherapy without piroxicam
  Arms: Mesotherapy without piroxicam and lidocaine

SUMMARY:
Investigate the short- and long-term efficacy and safety of intradermal NSAIDs and lidocaine (delivered through mesotherapy) for the treatment of LE comparing it with empty intradermal injections.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis defined as pain over the lateral epicondyle provoked by palpation;
* A visual analogue scale (VAS) score for pain greater than 40mm;
* symptoms duration for more than 1 month.

Exclusion Criteria:

* other diseases that can alter clinical evaluation detected through history, clinical examination, ultrasound or other exams for comorbidities such as carpal tunnel syndrome, cervical radiculopathy, elbow arthritis, intra-articular loose bodies, previous elbow surgery or clinically significant or recent trauma, fibromyalgia and major psychiatric conditions;
* VAS score for pain less than 40mm;
* any of the following treatments during the previous 4 weeks before baseline visit: physical therapy, bandage, mesotherapy and local corticosteroid injection or a combination of these: NSAIDS taken during the week previous to inclusion;
* pregnancy;
* allergy to any of the study drugs;
* severely immunosuppressed patients;
* known coagulopathies. During the study period, enrolled patients are not allowed to take oral corticosteroids, NSAIDs or receive any other medical intervention during the treatment period (physical therapy, bandage, mesotherapy and local corticosteroid injection or a combination of these).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-12 (Estimated); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: visual analogue scale score | 3 months
  pain intensity quantified by using a 0-100 visual analogue scale (VAS) score; a higher score means a higher pain intensity on the VAS

SECONDARY OUTCOMES:
Clinical and functional evaluation | 0, 1, 2, 3 weeks and 6 months
  American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES-E) score, ranging from 0 to 5 in strenght assessment (0=no contraction; 1=flicker; 2=movement with gravity eliminated; 3=movement against gravity; 4=movement with some resistance; 5=normal power) and from 0-3 in the stability section (0=no instability; 1=mild laxity with good endpoint; 2=moderate laxity no endpoint;3=gross instability)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided